CLINICAL TRIAL: NCT04989348
Title: A Randomized Control Trial to Compare the Euploid Rate of Blastocyst Between the Progestin-primed Ovarian Stimulation Protocol and the Gonadotrophin Releasing Hormone Antagonist Protocol in Patients With Undergoing Preimplantation Genetic Testing for Aneuploidy
Brief Title: Euploid Rate of Blastocyst Derived From PPOS VS Antagonist Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, chen zhi qin, clinical doctor in chief, Shanghai First Maternity and Infant Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: shanghaiFMIH-20210729
Record Dates: First submitted 2021-07-30; First posted 2021-08-04 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: IVF
Keywords: ppos; antagonist protocol; PGT-A; Euploid Rate of Blastocyst

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antagonist group (Placebo Comparator): Women will receive antagonist (Cetrorelix 0.25mg) once subcutaneously daily from day 6 of ovarian stimulation till the day of the ovulation trigger.
  Interventions: Procedure: Gonadotrophin releasing hormone antagonist protocol
- PPOS group (Active Comparator): Women will receive oral medroxyprogesterone 10 mg daily or Duphaston 10mg bd from Day 3 till the day of ovulation trigger.
  Gonadotrophin (human menopausal gonadotrophin or recombinant FSH) injections will be started. Ovarian response will be monitored by transvaginal scanning with or without serum hormonal level. Human chorionic gonadotrophin (hCG 1,000 IU) and GnRH agonist (decepepty 0.2mg) will be given for triggering of final maturation when at least 3 follicles reach >17mm in diameter. Blood will be checked for serum estradiol and progesterone levels. Transvaginal USS-guided oocyte retrieval will be performed 36 hours after the trigger.
  Interventions: Procedure: Progestin-primed ovarian stimulation protocol

INTERVENTIONS:
Procedure: Gonadotrophin releasing hormone antagonist protocol — Women will receive antagonist (Cetrorelix 0.25mg) once subcutaneously daily from day 6 of ovarian stimulation till the day of the ovulation trigger or
  Arms: Antagonist group
Procedure: Progestin-primed ovarian stimulation protocol — Women will receive oral medroxyprogesterone 10 mg daily or Duphaston 10mg bd from Day 3 till the day of ovulation trigger.
  Arms: PPOS group

SUMMARY:
In-vitro fertilization (IVF) involves multiple follicular development, oocyte retrieval and embryo transfer after fertilization. Despite recent advances in ovarian stimulation, the method of assisted fertilization and improved culture conditions, the implantation potential of embryos remains around 30-35% for a long time.

Gonadotrophin releasing hormone (GnRH) agonists have been used in IVF to prevent the LH surge and the premature ovulation and are given in the luteal phase of the preceding cycle or in the follicular phase of the treatment cycle i.e. the long GnRH agonist. GnRH antagonists are now commonly used during IVF. In addition to the advantage of its simplicity, the use of antagonist is associated with a substantial reduction in ovarian hyperstimulation syndrome without reducing the chance of achieving live birth when compared with the long agonist protocols. [1]

Progestin can inhibit the pituitary LH surge during ovarian stimulation and various studies show progestin-primed ovarian stimulation (PPOS) is effective in blocking the LH surge in IVF [2-5]. More and more centers in China are using PPOS because this regimen appears simpler and cheaper. Because of its negative effect on the endometrium, fresh transfer of embryos is not possible and elective freezing of all embryos is required. PPOS protocol is indicated in women who freeze all embryos because of various reasons such as undergoing preimplantation genetic testing for aneuploidy or the risk of ovarian hyperstimulation syndrome.

One prospective non-randomized study comparing the PPOS vs short GnRH agonist protocol shows similar oocytes retrieved between the two protocols, and the incidence of premature LH surge, clinical pregnancy rate and live birth rates shows no significant difference. [2] A recent randomized trial comparing medroxyprogesterone and GnRH antagonist in an oocyte donation program showed a similar number of mature oocytes but reported lower ongoing pregnancy rate and live birth rate of recipients of oocyte donors who had received medroxyprogesterone in IVF [6]. However, the oocyte recipients in that trial were not randomized. Therefore, it is not possible to conclude the effect of progestin used in IVF on the pregnancy outcomes. It is possible that the PPOS protocol may have an adverse effect on the euploid rate of embryos, leading to a lower live birth rate.

DETAILED DESCRIPTION:
The inability to assess embryo quality and select those with the highest potential for implantation on the basis of morphology has led to the concept of preimplantation genetic testing for aneuploidy (PGT-A). PGT-A involves biopsy of a few cells from an embryo and assessment of the chromosome copy numbers. While PGT-A cannot create a healthy embryo or improve the health of an embryo, it provides a method of selecting embryos with a normal number of chromosomes for transfer. This in turn has the potential to increase the chance of having a healthy live birth and reduce the risk of miscarriage or an abnormal fetus caused by an abnormal number of chromosomes. Aneuploidy screening of all chromosomes is necessary to determine whether an embryo is chromosomally normal.

As the turnaround time of PGT-A with next generation sequencing is about a week, it is not possible to transfer blastocyst in the stimulated cycle. All blastocysts will be frozen post biopsy and the blastocysts with normal genetic makeup will be thawed and replaced in a subsequent menstrual cycle. Cryopreservation of blastocysts and replacing the frozen blastocysts after thawing in subsequent cycles become a common practice with vitrification as the cryopreservation method. A systematic review (7) of the clinical utility of PGT-A with comprehensive chromosome screening found that three small randomised controlled trials demonstrated benefit in young and good prognosis patients in terms of clinical pregnancy rates and the use of single embryo transfer.

This randomized trial aims to compare the euploid rate of blastocysts between PPOS and GnRH antagonist protocols in patients undergoing PGT-A.

ELIGIBILITY:
Inclusion Criteria:

1. Age of women <43 years at the time of ovarian stimulation for IVF
2. PGT-A indicated for advanced maternal age (>40 years), recurrent miscarriage (>=2 or 3 consecutive miscarriage and repeated implantation failure (>=4 embryos replaced or >=2 blastocysts replaced without success)

Exclusion Criteria:

1. Presence of a functional ovarian cyst with E2>100 pg/mL
2. use of donor eggs/sperm,
3. Presence of hydrosalpinx or endometrial polyp which is not surgically treated
4. moderate or severe endometriosis

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
euploid blastocyst formation rate | 2 months
  Euploid blastocysts per injected MII oocyte

SECONDARY OUTCOMES:
Number of mature oocytes | 1 month
  M2 oocytes
Number of blastocysts suitable for biopsy and freezing | 1 month
  blastocysts after extented culture
clinical pregnancy of the first FET | an average of 3 months
  presence of intrauterine gestational sac on ultrasound
implantation rate | an average of 3 months
  number of gestational sacs per embryo transferred
ongoing pregnancy of the first FET | an average of 6 months
  viable pregnancy beyond gestation 10 weeks
live birth rate of the first FET | average of 1 year
  A baby born alive after 22 weeks gestation
Serum FSH level | 1 month
  hormone level
Serum AMH level | 1 month
  hormone level
Serum estradiol level | 1 month
  hormone level
Serum progesterone level | 1 month
  hormone level
incidence of premature LH surge | 1 month
  LH ≥10 IU/l

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai first Maternity and Infant health hospital, Tong Ji University, Shanghai, China

REFERENCES:
- [Result] Al-Inany HG, Youssef MA, Aboulghar M, Broekmans F, Sterrenburg M, Smit J, Abou-Setta AM. Gonadotrophin-releasing hormone antagonists for assisted reproductive technology. Cochrane Database Syst Rev. 2011 May 11;(5):CD001750. doi: 10.1002/14651858.CD001750.pub3. PMID 21563131
- [Result] Kuang Y, Chen Q, Fu Y, Wang Y, Hong Q, Lyu Q, Ai A, Shoham Z. Medroxyprogesterone acetate is an effective oral alternative for preventing premature luteinizing hormone surges in women undergoing controlled ovarian hyperstimulation for in vitro fertilization. Fertil Steril. 2015 Jul;104(1):62-70.e3. doi: 10.1016/j.fertnstert.2015.03.022. Epub 2015 May 5. PMID 25956370
- [Result] Dong J, Wang Y, Chai WR, Hong QQ, Wang NL, Sun LH, Long H, Wang L, Tian H, Lyu QF, Lu XF, Chen QJ, Kuang YP. The pregnancy outcome of progestin-primed ovarian stimulation using 4 versus 10 mg of medroxyprogesterone acetate per day in infertile women undergoing in vitro fertilisation: a randomised controlled trial. BJOG. 2017 Jun;124(7):1048-1055. doi: 10.1111/1471-0528.14622. PMID 28276192
- [Result] Massin N. New stimulation regimens: endogenous and exogenous progesterone use to block the LH surge during ovarian stimulation for IVF. Hum Reprod Update. 2017 Mar 1;23(2):211-220. doi: 10.1093/humupd/dmw047. PMID 28062551
- [Result] Yu S, Long H, Chang HY, Liu Y, Gao H, Zhu J, Quan X, Lyu Q, Kuang Y, Ai A. New application of dydrogesterone as a part of a progestin-primed ovarian stimulation protocol for IVF: a randomized controlled trial including 516 first IVF/ICSI cycles. Hum Reprod. 2018 Feb 1;33(2):229-237. doi: 10.1093/humrep/dex367. PMID 29300975
- [Result] Begueria R, Garcia D, Vassena R, Rodriguez A. Medroxyprogesterone acetate versus ganirelix in oocyte donation: a randomized controlled trial. Hum Reprod. 2019 May 1;34(5):872-880. doi: 10.1093/humrep/dez034. PMID 30927417
- [Result] Lee E, Illingworth P, Wilton L, Chambers GM. The clinical effectiveness of preimplantation genetic diagnosis for aneuploidy in all 24 chromosomes (PGD-A): systematic review. Hum Reprod. 2015 Feb;30(2):473-83. doi: 10.1093/humrep/deu303. Epub 2014 Nov 28. PMID 25432917
- [Derived] Wang L, Wang JY, Zhang Y, Qian C, Wang XH, Ng EHY, Ai A, Chen ZQ. Comparison of the euploidy rate in preimplantation genetic testing for aneuploidy cycles following progestin-primed versus gonadotropin-releasing hormone antagonist protocol: a randomized controlled study. Reprod Biol Endocrinol. 2025 May 13;23(1):67. doi: 10.1186/s12958-025-01404-0. PMID 40361159